CLINICAL TRIAL: NCT06094387
Title: The Use of Thrombin Generation Assay in Detection of Central Line Related Thrombosis (CRT) in Critically Ill Patients
Acronym: THROM-CRIT
Status: Recruiting | Type: Observational
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Wincy Wing-Sze Ng, Associate Consultant, Adult Intensive Care Unit, Queen Mary Hospital, Hong Kong
Other Study IDs: 20230905-017-000
Record Dates: First submitted 2023-10-13; First posted 2023-10-23 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Central Line Complication; Thrombosis, Venous
Keywords: Thrombin generation; Central line related thrombosis
MeSH Terms: conditions — Venous Thrombosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Thrombin generation assay — Thrombin generation parameters in patients receiving central catheter insertion

SUMMARY:
To study thrombin generation parameters in critically ill patients with and without central line related thrombosis (CRT).

ELIGIBILITY:
Inclusion Criteria:

* Age ≧ 18; AND
* Admitted to the mixed medical-surgical intensive care units of Queen Mary Hospital in Hong Kong; AND
* Clinically indicated for central catheter insertion, which includes central venous catheters and dialysis catheters; AND
* Expected to have the central catheter in place for at least 5 days in their ICU stay.

Exclusion Criteria:

* Patients known to have active venous thromboembolism including deep venous thrombosis or pulmonary embolism;
* Patients known to have hypercoagulable states, e.g., hereditary thrombophilia, antiphospholipid syndrome; OR
* Patients with active solid organ or hematological malignancies; OR
* Patients already receiving therapeutic anticoagulation prior to study recruitment; OR
* Patients with thrombosis detected in the insertion site before central catheter insertion; OR
* Patients with a central venous catheter already in place prior to ICU admission; OR
* Patients admitted to the ICU for post-operative care; OR
* Patients admitted to the ICU for trauma care; OR
* Patients requiring extra-corporeal life support (ECLS); OR
* Patients with poor window or inaccessible for ultrasonographic examination; OR
* Pregnancy/post-partum within 6 weeks

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients requiring central catheter insertion in the ICU
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-06 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Difference in peak thrombin generation (nM) between patients with and without central line related thrombosis | From the time of CVC insertion to the time of CVC removal
  The primary outcome measure is the difference in peak thrombin generation (nM) between patients with and without central line related thrombosis

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided